CLINICAL TRIAL: NCT00118872
Title: Feasibility Study of Probiotics for Growth Faltering in Pakistan
Brief Title: Beneficial Bacteria to Prevent Malnutrition and Diarrhea in Pakistani Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21AT001486-01A2 (NIH); R21AT001486 (NIH); Wanke 01
Record Dates: First submitted 2005-07-07; First posted 2005-07-12 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Malnutrition; Diarrhea
Keywords: Growth and Development; Pakistan; Weaning; Probiotics; Infant; Lactobacillus GG
MeSH Terms: conditions — Malnutrition; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LGG yogurt (Active Comparator): Lactobacillus (LGG) containing yogurt
  Interventions: Drug: LGG yogurt; Other: Placebo yogurt
- Placebo yogurt (Placebo Comparator): Regular yogurt, NOT containing LGG
  Interventions: Other: Placebo yogurt

INTERVENTIONS:
Drug: LGG yogurt — Lactobacillus GG containing yogurt
  Other Names: Lactobacillus GG containing yogurt
  Arms: LGG yogurt
Other: Placebo yogurt — Yogurt NOT containing the active LGG bacteria

SUMMARY:
This study will determine whether lactobacillus GG (LGG), a beneficial bacterium, when given in yogurt, will reduce growth faltering in babies living in a poor area of Pakistan who are being weaned from breastfeeding.

Study hypothesis: Use of the probiotic bacteria LGG at the time of weaning will lessen the impact of faltering growth in babies living in the slums of Pakistan.

DETAILED DESCRIPTION:
Faltering growth due to malnutrition and recurrent diarrhea is a serious public health concern in developing nations, particularly among infants who are being weaned from breastfeeding. Evidence suggests that the use of the probiotic bacterium LGG reduces the risk of diarrhea, shortens episodes of diarrhea, and enhances the immune system. Babies who are being weaned from breastfeeding will be given LGG-containing yogurt in this study to determine whether LGG will reduce faltering growth caused by diarrhea and malnutrition.

Infant participants will be enrolled at or within 5 weeks of birth and followed throughout the weaning period. During the weaning period, participants will be randomly assigned to either receive LGG-containing yogurt or placebo yogurt everyday for 3 months. All participants will have height and weight measurements taken at study entry and at Month 3 (study completion). The number of diarrhea episodes experienced by participants during the study will be assessed at study completion to determine participants' health.

ELIGIBILITY:
Inclusion Criteria:

* Born and reside in Bilal Colony, Karachi Pakistan during the study
* Parent or guardian willing to provide informed consent
* Parent or guardian willing to permit home visits
* Predominantly breastfed at study start

Exclusion Criteria:

* Malnutrition at time of weaning
* Medical condition that would affect response to LGG

Ages: 1 Week to 5 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Growth, as measured by weight for age and height | 3 months

SECONDARY OUTCOMES:
Number of episodes of diarrhea | 3 months
duration of episodes of diarrhea | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine A. Wanke, MD, Principal Investigator — Tufts University
Locations (1):
- Aga Khan Medical Center, Karachi, Pakistan